CLINICAL TRIAL: NCT01911559
Title: Effectiveness of Standing Frame on Constipation in Children With Cerebral Palsy: a Single Subject Study
Brief Title: Effectiveness of Standing Frame on Constipation in Children With Cerebral Palsy
Acronym: CP
Status: Completed | Type: Observational
Sponsor: Stefania Costi (Other)
Collaborators: Azienda Unita' Sanitaria Locale Di Modena (Other)
Responsible Party: Sponsor-Investigator, Stefania Costi, MSc in PT, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Other Study IDs: standing_2013
Record Dates: First submitted 2013-07-19; First posted 2013-07-30 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Palsy; Quadriplegia; Diplegia; Constipation
Keywords: Standing-frame; Chronic constipation; Cerebral palsy; Quadriplegia; Severe diplegia
MeSH Terms: conditions — Cerebral Palsy; Quadriplegia; Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- constipated quadriplegic CP children: In this study we included children with CP, in the manifestation of severe diplegia or quadriplegia, who do not currently use the standing-frame.
  Interventions: Device: standing-frame

INTERVENTIONS:
Device: standing-frame
  Other Names: stander

SUMMARY:
Children with Cerebral Palsy and quadriplegia or severe diplegia suffer from highly reduced mobility and consequent constipation. Clinicians frequently recommend standing-frames to exercise the support reaction in this population, sharing the opinion that the upright position may facilitate intestinal transit, although no evidence supports this assumption.

The investigators conducted this single-subject research to determine the effects of the standing-frame on the frequency of evacuation in chronically constipated children with CP and quadriplegia.

Moreover, the investigators studied its effects on the frequency of induction of evacuation, the characteristics of the stool and the pain suffered by the child due to constipation and/or evacuation.

ELIGIBILITY:
Inclusion criteria were:

* clinical indication for the use of the standing-frame;
* constipation problems as defined by guidelines (Clinical Practice Guideline, 2006);
* whose parents gave the informed consent to let their child to participate in this study.

Exclusion criteria were:

* children who have orthosympathetic reactions to the upright position, skeletal deformities and/or medical conditions that, according to clinical judgment, advise against the use of the standing frame.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In this study we included children with CP, in the manifestation of severe diplegia or quadriplegia, who do not currently use the standing-frame. The population of interest might be referred to the Unit for severe disability in developmental age or to one of the neuro-psychiatric and rehabilitation Units of the area of Modena and Reggio Emilia, (5.000 km2 of surface and 1.250.000 inhabitants)
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
bowel evacuation frequency | 14 weeks
  Using a daily-diary where the caregivers collect the data about the bowel evacuation frequency

SECONDARY OUTCOMES:
Bowel evacuation inductions frequency | 14 weeks
  Using a daily-diary where the caregivers collect the data about the bowel evacuation inductions frequency

OTHER OUTCOMES:
pain related to the bowel evacuation | 14 weeks
  Using a daily-diary where the caregivers collect the data about the pain related to the bowel evacuation
distress of the caregiver | 14 weeks
  Using a daily-diary where the caregivers collect the data about the distress of the caregiver

CONTACTS AND LOCATIONS:
Locations (1):
- Local Health Institution of Modena, Carpi, Modena, Italy

REFERENCES:
- [Background] Pin TW. Effectiveness of static weight-bearing exercises in children with cerebral palsy. Pediatr Phys Ther. 2007 Spring;19(1):62-73. doi: 10.1097/PEP.0b013e3180302111. PMID 17304099
- Available data/document: Clinical Study Report: 9433361 — http://www.biomedsearch.com/nih/Effectiveness-Standing-Frame-Constipation-in/24838311.html — Rivi, Elena & Filippi, Mariacristina & Fornasari, Elisa & Mascia, Maria Teresa & Ferrari, Adriano & Costi, Stefania. (2014). Effectiveness of Standing Frame on Constipation in Children with Cerebral Palsy: A Single-Subject Study. Occupational therapy international.